CLINICAL TRIAL: NCT05371002
Title: Effectiveness of Online Group-based Nonviolent Communication Interventions for Reducing Parenting Stress in Parents With Mild to Moderate Depressive Symptoms: a Randomized Controlled Trial
Brief Title: Effectiveness of Online Group-based Nonviolent Communication Interventions
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to lack of funding source, the main trial has been suspended. The research team is looking for funding source to recover the trial.
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Yuying Sun, Research Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 17605422
Record Dates: First submitted 2022-05-03; First posted 2022-05-12 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Mild to Moderate Depressive Symptoms
Keywords: depression; parents
MeSH Terms: conditions — Depression | interventions — Methods

STUDY DESIGN:
Intervention Model Description: A parallel individual RCT with two groups: (1) an intervention group receiving online group based NVC training and (2) a waitlist control (WL) group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Online group nonviolent communication (NVC) interventions (Experimental): Rosenberg's "Nonviolent Communication: A Language of Life: Life-changing Tools for Healthy Relationships" and "Raising Children Compassionately: Parenting the Nonviolent Communication Way" will be used as reference guides. Six 1.5-hour weekly online group sessions (10-14 participants in each group) will be delivered by NVC professionals to the intervention group, including (1) introduction to four key principles of NVC, communication that blocks compassion, and distinguishing observations from evaluations, (2) identifying and expressing feelings, providing a list of words to express feelings and four steps to express anger, (3) taking responsibility for feelings (needs), distinguishing between an outside event and the met or unmet needs behind the feelings, (4) using positive action language to make requests, (5) review and summary, and (6) experience sharing and suggestions for further practice. Group discussion will be used to sustain the participants' engagement.
  Interventions: Behavioral: Online group nonviolent communication (NVC) interventions
- Waitlist control group (Active Comparator): The participants in WL group will not be provided any materials or training content between baseline (T1) and immediate post assessment (T2). Once the participants completed the T2 assessments, they will be delivered one 1.5-hour online session about physical activity (completely different from NVC training content). In the session, the participants will be introduced the concept of Zero-time exercise and provided video demonstrations of exercise. Six 1.5-hour weekly NVC training sessions (the same as those in intervention group) will be delivered to participants as soon as they have completed the final assessment at T3 (three months after T2).
  Interventions: Other: Waitlist control group

INTERVENTIONS:
Behavioral: Online group nonviolent communication (NVC) interventions — The primary purpose of NVC as defined by Dr. Marshall Rosenberg is to resolve interpersonal conflict using empathic communication skills. Nonviolence does not refer to the mere absence of physical harm. It is a way of life that helps us to transform old patterns of defensiveness and aggressiveness into compassion and empathy and to improve the quality of all types of relationships. The basic model of NVC consists of four key principles: the separation of observation from evaluation (observation), exploring and expressing the feelings that emerge from observations (feeling), taking responsibility for one's feelings (need), and telling others the need to enrich lives (request). A book on NVC specifically targets parents to improve communication and connection with their children. The NVC model emphasizes the importance of observation and has similarities with the concept of "mindful parenting", which refers to a non-judgmental and open parenting style.
  Arms: Online group nonviolent communication (NVC) interventions
Other: Waitlist control group — Waitlist control, but included a short active intervention during the 2nd and 3rd assessments.
  Arms: Waitlist control group

SUMMARY:
This is a randomized controlled trial (RCT) to test the effectiveness of nonviolent communication (NVC) intervention for reducing parenting stress to parents with children in primary schools and mild to moderate depression. A pilot RCT on 50 participants (25 in NVC vs. 25 in control group, 2 small groups for each arm) will be conducted in late June to September 2022 to test the procedure and preliminary results. A RCT (1:1 allocation ratio) on 200 parents who have children of Grade 1-6 and mild to moderate depressive symptoms assessed by Patient Health Questionnaire (PHQ)-9. Outcomes will be measured at baseline, immediately after completion of intervention and three months after the intervention. This study will provide evidence on the effectiveness of NVC to reduce parenting stress and enhance parents' mental well-being.

DETAILED DESCRIPTION:
Objectives: To test the effectiveness of nonviolent communication (NVC) intervention for reducing parenting stress in parents with mild to moderate depression and children in primary schools.

Hypothesis: Our intervention group will show more improvements in parents' NVC skills, parenting stress, depression and anxiety symptoms, and well-being than the control group.

Design and subjects: An RCT (1:1 allocation ratio) on 200 parents who have mild to moderate depressive symptoms assessed by Patient Health Questionnaire (PHQ)-9 and children of Grade 1-6.

Instruments: Parental Stress Scale; self-developed NVC scale; PHQ-9; Generalized Anxiety Disorder-7; Short Warwick-Edinburgh Mental Well-being Scale.

Interventions: Six 1.5-hour weekly online group sessions (10-14 participants in each group) will be delivered by NVC professionals to the intervention group, including (1) introduction to four key principles of NVC, communication that blocks compassion, and distinguishing observations from evaluations, (2) identifying and expressing feelings, providing a list of words to express feelings and four steps to express anger, (3) taking responsibility for feelings (needs), distinguishing between an outside event and the met or unmet needs behind the feelings, (4) using positive action language to make requests, (5) review and summary, and (6) experience sharing and suggestions for further practice. Group discussion will be used to sustain the participants' engagement. The waitlist control group will receive simple messages through the same media on physical activity and will be provided with the training sessions afterwards. A pilot study on 50 participants (25 in NVC vs. 25 in control group, 2 small groups for each arm) will be conducted in late June to September 2022 to test the procedure and preliminary results. Only T1 and T2 will be conducted to obtain the immediate effect of the intervention.

Outcome measures: Outcomes will be measured at baseline, immediately after completion of intervention and three months after the intervention. The primary outcome is parenting stress at 3-month after the intervention. Secondary outcomes include NVC skills, parental depression and anxiety symptoms, and well-being at 3-month after the intervention. Process evaluation will be conducted after the intervention. In-depth interviews will be conducted on 30 parents in the intervention group to explore participants' experiences.

Data analysis: Intention-to-treat approach. A multilevel mixed model will be used to evaluate the between-group mean differences in the outcomes of the two groups, after adjusting for baseline outcomes and demographics. Per-protocol sensitivity analyses will be conducted by only including the adherent participants who complete at least four sessions and all assessments. Mediation analysis will be conducted following AGReMA guideline. Cost analysis will be conducted.

Expected results: The intervention group will show greater improvements in the measured outcomes than the control group, offering strong evidence of effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* Parents with children in primary schools (Grade 1-6, age 6-12), aged 24-59 years;
* With mild to moderate depressive symptoms (score of 5-14 on the PHQ-9);
* Hong Kong residents who can communicate in Chinese (Cantonese or Mandarin).

Exclusion Criteria:

* Have been diagnosed as major depressive disorder in the past 6 months;
* Under psychiatric treatment;
* Currently participating in other parenting or related programs;
* Parents with PHQ score > 14 will be advised to consult a doctor.

Ages: 24 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 250 (Estimated)
Dates: Start 2022-05-16 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Changes in parenting stress | T1: baseline; T2: immediate post-intervention; T3: 3-month after the intervention
  Parenting stress will be assessed by Parental Stress Scale (PSS). An 16-item PSS has been developed by Leung et al for Hong Kong Chinese parents. It assesses the parenting stress using a 5-point response scale, ranging from 18 to 80.

SECONDARY OUTCOMES:
Changes in NVC skills | T1: baseline; T2: immediate post-intervention; T3: 3-month after the intervention
  A Chinese version will be developed based on the four core components of NVC, with each item rated on a 5-point scale ranging from 0 = never to 5 = always. The average score will be calculated, with higher scores indicating better NVC skills.
Changes in depressive symptoms | T1: baseline; T2: immediate post-intervention; T3: 3-month after the intervention
  The Patient Health Questionnaire (PHQ)-9 will be used to measure depressive symptoms. Participants rate the frequency of nine symptoms over the past two weeks on a 4-point Likert scale (from 0=not at all to 3=nearly every day). The total score ranges from 0 to 27, with higher scores indicating a greater severity of depressive symptoms.
Changes in anxiety symptoms | T1: baseline; T2: immediate post-intervention; T3: 3-month after the intervention
  Generalized Anxiety Disorder (GAD)-7 will be used to assess generalized anxiety disorder. Participants rate the frequency of seven symptoms over the past two weeks on a 4-point Likert scale (from 0=not at all to 3=nearly every day). The total score ranges from 0 to 21, with a higher score indicating a higher level of anxiety.
Changes in well-being | T1: baseline; T2: immediate post-intervention; T3: 3-month after the intervention
  The 7-item Short Warwick-Edinburgh Mental Well-being Scale with the 5-point Likert scale (1 = none of the time, 5 = all the time) will be used. The score is calculated by summing all seven items with a range of 7 to 35. A higher score indicated higher level of wellbeing.

OTHER OUTCOMES:
Subjective changes in personal mental health | T2: immediate post-intervention; T3: 3-month after the intervention
  The subjective changes in personal mental health compared with baseline will be rated on 5-point Likert scale, with "5" indicating "much better", "3" indicated "no change" and "1" indicated "much worse".
Subjective changes in parent-child conflict | T2: immediate post-intervention; T3: 3-month after the intervention
  The subjective changes in parent-child conflict compared with baseline will be rated on 5-point Likert scale, with "5" indicating "much better", "3" indicated "no change" and "1" indicated "much worse".
Subjective changes in parent-child communication | T2: immediate post-intervention; T3: 3-month after the intervention
  The subjective changes in parent-child communication compared with baseline will be rated on 5-point Likert scale, with "5" indicating "much better", "3" indicated "no change" and "1" indicated "much worse".
The overall satisfaction with the NVC courses | T2: immediate post-intervention; T3: 3-month after the intervention
  The overall satisfaction with the NVC courses will be rated on a 0-10 scale by the participants, with "0" indicating "very unsatisfied" and "10" indicating "very satisfied".

CONTACTS AND LOCATIONS:
Overall Officials: Yuying Sun, PhD, Principal Investigator — School of Public Health, The University of Hong Kong
Locations (1):
- School of Nursing and Health Studies, Hong Kong Metropolitan University, Hong Kong, China